CLINICAL TRIAL: NCT00050778
Title: A Phase II, Randomized, Open-Label, Three-Arm Study Comparing Low- and High-Dose Alemtuzumab and High-Dose Subcutaneous Interferon Beta-1a (Rebif®) in Patients With Early, Active Relapsing-Remitting Multiple Sclerosis
Brief Title: A Phase II Study Comparing Low- and High-Dose Alemtuzumab and High-Dose Rebif® in Patients With Early, Active Relapsing-Remitting Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CAMMS223
Record Dates: First submitted 2002-12-19; First posted 2002-12-23 (Estimated); Results first posted 2009-08-25 (Estimated); Last update posted 2015-01-08 (Estimated); Status verified 2015-01

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Active Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1a; Alemtuzumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interferon Beta-1a (Active Comparator)
  Interventions: Biological: Interferon beta-1a
- Alemtuzumab 12 mg (Experimental)
  Interventions: Biological: Alemtuzumab 12 mg
- Alemtuzumab 24 mg (Experimental)
  Interventions: Biological: Alemtuzumab 24 mg

INTERVENTIONS:
Biological: Interferon beta-1a — Interferon beta-1a 44 microgram (mcg) subcutaneously 3-times weekly for 36 months.
  Other Names: Rebif®
  Arms: Interferon Beta-1a
Biological: Alemtuzumab 12 mg — Alemtuzumab 12 milligram per day (mg/day) was given by intravenous infusion on 5 consecutive days during the first month and on 3 consecutive days at months 12 and 24 (the latter at the treating physicians' discretion if the cluster of differentiation 4+ [CD4+] T-cell count was >=100*10^6 cells per liter).
  Other Names: Lemtrada
  Arms: Alemtuzumab 12 mg
Biological: Alemtuzumab 24 mg — Alemtuzumab 24 mg/day was given by intravenous infusion on 5 consecutive days during the first month and on 3 consecutive days at months 12 and 24 (the latter at the treating physicians' discretion if the CD4+ T-cell count was >=100*10^6 cells per liter).
  Other Names: Lemtrada
  Arms: Alemtuzumab 24 mg

SUMMARY:
This was a Phase II, randomized, open-label, rater-blinded, three-arm study comparing two different doses of alemtuzumab (Lemtrada™) and one dose of subcutaneous (SC) interferon beta-1a (Rebif®) in participants with early, active relapsing-remitting multiple sclerosis (MS) who had not been previously treated with MS therapies other than steroids. The study was conducted for an initial period of 3 years and a follow-up to 5 years or more.

DETAILED DESCRIPTION:
The aims of MS therapy are to prevent the progression of disease and accumulation of long-term disability. The hypothesis underlying this study was that aggressive treatment of inflammation in the brain early in the course of MS would protect the participant from disease progression and accumulating disability.

This protocol compared two different doses of alemtuzumab and high-dose, high frequency of SC interferon beta-1a to evaluate the safety profiles of the respective treatments and to evaluate efficacy in terms of:

* Slowing the sustained accumulation of disability in participant with MS;
* Reducing the frequency of relapses experienced by participant with MS; and
* Reducing the harmful effects of MS on the brain, as assessed by magnetic resonance imaging (MRI)

Participants who received alemtuzumab during the initial 36-month treatment period may have been eligible for re-treatment with alemtuzumab in the extension study CAMMS03409 (NCT00930553) to evaluate:

* How long the effects of prior alemtuzumab treatment lasted;
* If additional treatments with alemtuzumab continued to reduce the effects of MS; and
* What kind of side effects participants experienced upon retreatment with alemtuzumab

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Male or non-pregnant, non-lactating female participants, 18 to 50 years of age (inclusive) as of signing the ICF
* Diagnosis of MS per McDonald's update of the Poser criteria, including cranial MRI consistent with those criteria (McDonald, 2001, Ann Neurol)
* Onset of first MS symptoms within 3 years prior to Screening as of signing the ICF
* Expanded Disability Status Scale (EDSS) score 0.0 to 3.0 (inclusive) at the screening and Baseline visits
* At least 2 completed clinical episodes of MS in the 2 years prior to study entry (that is, the initial event if within 2 years of study entry plus at least 1 relapse, or at least 2 relapses if the initial event was between 2 and 3 years prior to study entry)
* In addition to the clinical criteria, at least 1 enhancing lesion on any 1 of up to 4 screening gadolinium-enhanced MRI brain scans during a maximum 3-month run-in period (inclusive of the Month 0 Baseline scan)

Exclusion Criteria:

* Previous immunotherapy for MS other than steroids, including treatment with interferons, intravenous immunoglobulin (IVIG), glatiramer acetate, and mitoxantrone
* Personal history of thyroid autoimmune disease
* Personal history of clinically significant autoimmune disease (for example, inflammatory bowel disease, diabetes, lupus, severe asthma)
* History of thyroid carcinoma (previous thyroid adenoma was acceptable and was not considered an exclusion criterion)
* History of malignancy (except for basal cell skin carcinoma if disease-free for at least 5 years)
* Any disability acquired from trauma or another illness that, in the opinion of the Investigator, interfered with evaluation of disability due to MS
* Previous treatment with alemtuzumab
* History of anaphylaxis following exposure to humanized monoclonal antibodies
* Inability to undergo MRI with gadolinium administration
* Female participants of childbearing potential with a positive serum pregnancy test at screening or Baseline
* Male and female participants who did not agree to use effective contraceptive method(s) during the study
* Impaired renal function (that is, serum creatinine greater than or equal to 2 times the upper limit of normal [ULN])
* Untreated, major depressive disorder
* Epileptic seizures that were not adequately controlled by treatment
* Suicidal ideation
* Major systemic disease or other illness that, in the opinion of the Investigator, have compromised participant safety or interfered with the interpretation of study results
* Abnormal CD4 count or significantly abnormal thyroid function; presence of anti-thyroid stimulating hormone (TSH) receptor antibodies; known seropositivity for human immunodeficiency (HIV)
* Intolerance of pulsed corticosteroids, especially a history of steroid psychosis
* Presence of a monoclonal paraprotein
* Participants who had any form of MS other than relapsing-remitting
* Participants currently participating in a clinical study of an experimental or unapproved/unlicensed therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 334 (Actual)
Dates: Start 2002-12; Primary Completion 2007-09 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (49):
- United States (31):
  - Mayo Clinic Scottsdale Arizona, Scottsdale, Arizona
  - Clinical Trials, Inc, Little Rock, Arkansas
  - East Bay Physicians Medical Group, Berkeley, California
  - Nerve Pro Research, Irvine, California
  - Neuro-Therapeutics, Inc., Pasadena, California
  - Neurological Research Institute of the East Bay, Walnut Creek, California
  - Neurologic Research Institute/Mile High Research Center, Denver, Colorado
  - Neurological Service of Orlando, Orlando, Florida
  - Neurological Associates/ Research Dept., Pompano Beach, Florida
  - Neurology Clinical Research, Inc., Sunrise, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Medical Research and Health Education, Columbus, Georgia
  - Consultants in Neurology, Ltd, Northbrook, Illinois
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Associate in Neurology, Lexington, Kentucky
  - University of Maryland -Maryland Center for MS, Baltimore, Maryland
  - Wayne State University Department of Neurology, Detroit, Michigan
  - Michigan Institute for Neurological Disorders, Farmington Hills, Michigan
  - Michigan Medical P.C. Neurology, Grand Rapids, Michigan
  - Mayo Clinic Rochester Department of Neurology, Rochester, Minnesota
  - Nevada Neurological Consultants, Ltd., Las Vegas, Nevada
  - University Hospital an Medical Center, Stony Brook, New York
  - ALL-Trials Clinical Research, LLC, Winston-Salem, North Carolina
  - Neurological Associates of Tulsa, Inc, Tulsa, Oklahoma
  - Neurosciencies and Pain Research, Allentown, Pennsylvania
  - Neurology, PC, Knoxville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Dallas Neurological Associate, Richardson, Texas
  - Central Texas Neurology Consultants PA, Round Rock, Texas
  - Integra Clinical Research, LLC, San Antonio, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
- Croatia (5):
  - Department of Neurology, University Hospital "Osijek", Osijek
  - Department of Neurology, Clinical Hospital Centre "Rijeka", Rijeka
  - Department of Neurology, Clinical Hospital Centre "Zagreb", Zagreb
  - Department of Neurology, General Hospital "Sveti Duh", Zagreb
  - Department of Neurology, University Hopsital "Sestre Milosrdnice", Zagreb
- Poland (6):
  - Centrum Neurologii Klinicznej, Krakow
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej, Lodz
  - Klinika Neurologii, Lublin
  - Oddzial Kliniczny Neurologii, Poznan
  - Instytut Psychiatrii i Neurologii, Warsaw
  - Katedra i Klinika Neurologii, Warsaw
- Russia (6):
  - Russian State Medical University, Moscow
  - Neurology Scientific Center RAMS, Moscow
  - Moscow City Hospital #11, Moscow
  - Moscow City Hospital #61, Moscow
  - Institute of Human brain RAS, Saint Petersburg
  - St. Petersburg State Pavlov Medical University, Saint Petersburg
- Addenbrooke's Hospital, Cambridge, England, United Kingdom

REFERENCES:
- [Background] Coles AJ, Cox A, Le Page E, Jones J, Trip SA, Deans J, Seaman S, Miller DH, Hale G, Waldmann H, Compston DA. The window of therapeutic opportunity in multiple sclerosis: evidence from monoclonal antibody therapy. J Neurol. 2006 Jan;253(1):98-108. doi: 10.1007/s00415-005-0934-5. Epub 2005 Jul 27. PMID 16044212
- [Result] CAMMS223 Trial Investigators; Coles AJ, Compston DA, Selmaj KW, Lake SL, Moran S, Margolin DH, Norris K, Tandon PK. Alemtuzumab vs. interferon beta-1a in early multiple sclerosis. N Engl J Med. 2008 Oct 23;359(17):1786-801. doi: 10.1056/NEJMoa0802670. PMID 18946064
- [Result] Daniels GH, Vladic A, Brinar V, Zavalishin I, Valente W, Oyuela P, Palmer J, Margolin DH, Hollenstein J. Alemtuzumab-related thyroid dysfunction in a phase 2 trial of patients with relapsing-remitting multiple sclerosis. J Clin Endocrinol Metab. 2014 Jan;99(1):80-9. doi: 10.1210/jc.2013-2201. Epub 2013 Dec 20. PMID 24170099
- [Result] Graves J, Galetta SL, Palmer J, Margolin DH, Rizzo M, Bilbruck J, Balcer LJ. Alemtuzumab improves contrast sensitivity in patients with relapsing-remitting multiple sclerosis. Mult Scler. 2013 Sep;19(10):1302-9. doi: 10.1177/1352458513475722. Epub 2013 Mar 4. PMID 23459567
- [Result] Coles AJ, Fox E, Vladic A, Gazda SK, Brinar V, Selmaj KW, Skoromets A, Stolyarov I, Bass A, Sullivan H, Margolin DH, Lake SL, Moran S, Palmer J, Smith MS, Compston DA. Alemtuzumab more effective than interferon beta-1a at 5-year follow-up of CAMMS223 clinical trial. Neurology. 2012 Apr 3;78(14):1069-78. doi: 10.1212/WNL.0b013e31824e8ee7. Epub 2012 Mar 21. PMID 22442431
- [Result] Coles AJ, Fox E, Vladic A, Gazda SK, Brinar V, Selmaj KW, Bass AD, Wynn DR, Margolin DH, Lake SL, Moran S, Palmer J, Smith MS, Compston DA. Alemtuzumab versus interferon beta-1a in early relapsing-remitting multiple sclerosis: post-hoc and subset analyses of clinical efficacy outcomes. Lancet Neurol. 2011 Apr;10(4):338-48. doi: 10.1016/S1474-4422(11)70020-5. PMID 21397567
- [Result] Jones JL, Anderson JM, Phuah CL, Fox EJ, Selmaj K, Margolin D, Lake SL, Palmer J, Thompson SJ, Wilkins A, Webber DJ, Compston DA, Coles AJ. Improvement in disability after alemtuzumab treatment of multiple sclerosis is associated with neuroprotective autoimmunity. Brain. 2010 Aug;133(Pt 8):2232-47. doi: 10.1093/brain/awq176. Epub 2010 Jul 21. PMID 20659956
- [Result] Cuker A, Coles AJ, Sullivan H, Fox E, Goldberg M, Oyuela P, Purvis A, Beardsley DS, Margolin DH. A distinctive form of immune thrombocytopenia in a phase 2 study of alemtuzumab for the treatment of relapsing-remitting multiple sclerosis. Blood. 2011 Dec 8;118(24):6299-305. doi: 10.1182/blood-2011-08-371138. Epub 2011 Sep 29. PMID 21960587
- [Derived] Riera R, Torloni MR, Martimbianco ALC, Pacheco RL. Alemtuzumab for multiple sclerosis. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD011203. doi: 10.1002/14651858.CD011203.pub3. PMID 37272540
- [Derived] Coles AJ, Jones JL, Vermersch P, Traboulsee A, Bass AD, Boster A, Chan A, Comi G, Fernandez O, Giovannoni G, Kubala Havrdova E, LaGanke C, Montalban X, Oreja-Guevara C, Piehl F, Wiendl H, Ziemssen T. Autoimmunity and long-term safety and efficacy of alemtuzumab for multiple sclerosis: Benefit/risk following review of trial and post-marketing data. Mult Scler. 2022 Apr;28(5):842-846. doi: 10.1177/13524585211061335. Epub 2021 Dec 9. PMID 34882037
- [Derived] Li Z, Richards S, Surks HK, Jacobs A, Panzara MA. Clinical pharmacology of alemtuzumab, an anti-CD52 immunomodulator, in multiple sclerosis. Clin Exp Immunol. 2018 Dec;194(3):295-314. doi: 10.1111/cei.13208. Epub 2018 Oct 1. PMID 30144037
- [Derived] Fox EJ, Wynn D, Coles AJ, Palmer J, Margolin DH; CAMMS223 Investigators. Alemtuzumab improves neurological functional systems in treatment-naive relapsing-remitting multiple sclerosis patients. J Neurol Sci. 2016 Apr 15;363:188-94. doi: 10.1016/j.jns.2016.02.025. Epub 2016 Feb 12. PMID 27000249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 49 investigational sites in the United States, United Kingdom, and Eastern Europe between December 04, 2002 and January 12, 2010.
Groups:
- Interferon Beta-1a: Interferon beta-1a (Rebif®) 44 micrograms (mcg) subcutaneously 3-times weekly for 36 months.
- Alemtuzumab 12 mg: Alemtuzumab (Lemtrada™) 12 milligram per day (mg/day) was given by intravenous infusion on 5 consecutive days during the first month and on 3 consecutive days at months 12 and 24 (the latter at the treating physicians' discretion if the cluster of differentiation 4+ [CD4+] T-cell count was >=100*10^6 cells per liter).
Period: Overall Study
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg
Started | 111 (Randomized.) | 113 | 110
Treated | 107 | 108 | 108
Completed | 66 | 92 | 92
Not Completed | 45 | 21 | 18
Not completed — Adverse Event | 13 | 3 | 2
Not completed — Death | 0 | 1 | 1
Not completed — Lack of Efficacy | 16 | 2 | 2
Not completed — Lost to Follow-up | 0 | 2 | 4
Not completed — Physician Decision | 3 | 0 | 2
Not completed — Protocol Violation | 2 | 0 | 1
Not completed — Withdrawal by Subject | 6 | 8 | 4
Not completed — Randomized but not treated | 4 | 5 | 2
Not completed — Familial and personal reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: FAS population included all randomized participants who had correct diagnosis of MS at entry. One participant was included in safety but excluded from efficacy analysis as initial multiple sclerosis diagnosis was incorrect.
Groups:
- Interferon Beta-1a: Interferon beta-1a 44 mcg subcutaneously 3-times weekly for 36 months.
- Alemtuzumab 12 mg: Alemtuzumab 12 mg/day was given by intravenous infusion on 5 consecutive days during the first month and on 3 consecutive days at months 12 and 24 (the latter at the treating physicians' discretion if the CD4+ T-cell count was >=100*10^6 cells per liter).
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Total
Number analyzed (Participants) | 111 | 112 | 110 | 333
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (8.82) | 31.9 (8.01) | 32.2 (8.76) | 32.3 (8.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 71 | 72 | 71 | 214
  Male | 40 | 40 | 39 | 119
Time Since First Relapse [Median (Full Range); unit: years] | 1.4 [0.2 to 6.3] | 1.3 [0.1 to 3.5] | 1.2 [0.3 to 3.2] | 1.3 [0.1 to 6.3]
Number of Relapse Episodes in the Preceding 2 Years [Number; unit: participants] — Number of participants with 0, 1, 2 or greater than or equal to 3 relapses are reported.
  participants
    0 Relapse | 0 | 2 | 1 | 3
    1 Relapse | 8 | 5 | 13 | 26
    2 Relapses | 73 | 58 | 56 | 187
    Greater than or equal to 3 Relapses | 30 | 47 | 40 | 117
Total Number of Relapses [Number; unit: relapses] | 293 | 301 | 290 | 884
Expanded Disability Status Scale (EDSS) Score [Mean (Standard Deviation); unit: units on a scale] — EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses the 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score ranges from 0 (normal neurological examination) to 10 (death due to MS). Number of participants evaluable for this Baseline characteristic were 110, 112 and 110 in Interferon Beta-1a, Alemtuzumab 12 mg and Alemtuzumab 24 mg arm, respectively.
  units on a scale | 1.9 (0.81) | 2.0 (0.73) | 2.0 (0.73) | 1.9 (0.76)
Time Constant 1 (T1) Cerebral Volume [Mean (Standard Deviation); unit: cubic centimeter] — Number of participants evaluable for this Baseline characteristic were 103, 107 and 107 in Interferon Beta-1a, Alemtuzumab 12 mg and Alemtuzumab 24 mg arm, respectively. Partial brain volumes were measured using the technique of Losseff et al. (1996).
  cubic centimeter | 317.5 (24.70) | 320.8 (27.15) | 320.5 (24.99) | 319.6 (25.61)
Time Constant 2 (T2) Lesion Volume [Mean (Standard Deviation); unit: cubic centimeter] — Number of participants evaluable for this Baseline characteristic were 102, 106 and 107 in Interferon Beta-1a, Alemtuzumab 12 mg and Alemtuzumab 24 mg arm, respectively.
  cubic centimeter | 15.8 (15.23) | 17.2 (23.84) | 17.8 (17.45) | 17.0 (19.19)

OUTCOME MEASURES:

1. Primary Outcome: Probability of Participants With Sustained Accumulation of Disability (SAD)
Description: EDSS is an ordinal scale in half-point increments that quantifies disability in participants with MS. It assesses 7 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder and cerebral) as well as ambulation. EDSS total score: 0 (normal neurological examination) to 10 (death due to MS). As measured by EDSS score, SAD was defined as increase of at least 1.5 points for participants with Baseline score of 0 and increase of at least 1.0 point for participants with Baseline score of 1.0 or more; and the increase persisted for at least next the 2 scheduled assessments, that is, 6 consecutive months. The onset date of SAD was date of first EDSS assessment that began 6 month consecutive period of SAD. Participants who did not reach SAD endpoint were censored at their last visit. Probability of participants with SAD, estimated by Kaplan-Meier (KM) method, was reported.
Time Frame: Up to 3 years
Population: Full Analysis Set (FAS) population included all randomized participants who had correct diagnosis of MS at entry.
Measure: Number (95% Confidence Interval); unit: probability of participants with SAD
Groups:
- Alemtuzumab (Pooled): Included all participants who received alemtuzumab 12 mg/day or 24 mg/day by intravenous infusion on 5 consecutive days during first month and on 3 consecutive days at months 12 and 24 (the latter at the treating physicians' discretion if the CD4+ T-cell count was >=100*10^6 cells per liter).
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Alemtuzumab (Pooled)
Number analyzed (Participants) | 111 | 112 | 110 | 222
probability of participants with SAD | 0.27 [0.193 to 0.380] | 0.08 [0.043 to 0.165] | 0.09 [0.052 to 0.169] | 0.09 [0.057 to 0.139]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Cox proportional hazards (PH) regression model using treatment group, Baseline EDSS group (grouped by less than or equal to 1.5 and greater than 1.5), and country (investigative center grouped by country) as covariates was used; Test type: Superiority or Other; p = 0.0006, Cox Proportional Hazards Regression — An alpha-sharing approach was used to adjust for multiple treatment group comparisons, endpoints, and two pre-planned interim analyses, including a Lan-Demets error-spending function. Pre-specified threshold for statistical significance was 0.0165; Hazard Ratio (HR) = 0.24, 95% CI 2-sided [0.110 to 0.545]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Alemtuzumab 24 mg; Cox PH regression model using treatment group, Baseline EDSS group (grouped by less than or equal to 1.5 and greater than 1.5), and country (investigative center grouped by country) as covariates was used; Test type: Superiority or Other; p = 0.0021, Cox Proportional Hazards Regression — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.151 to 0.658]
Statistical Analysis 3: Comparison: Interferon Beta-1a vs Alemtuzumab (Pooled); [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazards Regression; Hazard Ratio (HR) = 0.28, 95% CI 2-sided [0.152 to 0.515]

2. Primary Outcome: Annualized Relapse Rate
Description: Relapse was defined as new neurological symptoms or worsening of previous neurological symptoms with an objective change on neurological examination, attributable to multiple sclerosis that lasted for at least 48 hours, that were present at normal body temperature, and that were preceded by at least 30 days of clinical stability. Annualized relapse rate was estimated using a Poisson regression model with observed number of relapses as a dependent variable, the log total amount of follow-up from date of randomization for each participant as an offset variable and treatment group indicator as a covariate.
Time Frame: Up to 3 years
Population: FAS population included all randomized participants who had correct diagnosis of MS at entry.
Measure: Number (95% Confidence Interval); unit: relapses per participant per year
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Alemtuzumab (Pooled)
Number analyzed (Participants) | 111 | 112 | 110 | 222
relapses per participant per year | 0.37 [0.297 to 0.449] | 0.12 [0.091 to 0.171] | 0.09 [0.064 to 0.133] | 0.11 [0.085 to 0.137]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Treatment effects were estimated using an Anderson-Gill multiplicative intensity model with robust variance estimation. Covariates included treatment group, Baseline EDSS group (grouped by less than or equal to 1.5 and greater than 1.5), and country (investigative center grouped by country); Test type: Superiority or Other; p < 0.0001, Andersen-Gill Model — An alpha-sharing approach was used to adjust for multiple treatment group comparisons, endpoints, and two pre-planned interim analyses, including a Lan-Demets error-spending function. Pre-specified threshold for statistical significance was 0.0040; Rate ratio = 0.33, 95% CI 2-sided [0.196 to 0.552]
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Alemtuzumab 24 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Andersen-Gill Model — [p-value comment as in outcome 2, analysis 1]; Rate ratio = 0.23, 95% CI 2-sided [0.126 to 0.431]
Statistical Analysis 3: Comparison: Interferon Beta-1a vs Alemtuzumab (Pooled); [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Andersen-Gill Model; Rate ratio = 0.28, 95% CI 2-sided [0.176 to 0.441]

3. Secondary Outcome: Probability of Participants Who Were Relapse Free at 3 Years After Initial Treatment
Description: Participants were considered relapse free at Year 3 if they did not experience a relapse between randomization and study completion at 36 months. Participants who discontinued early were considered relapse free if they did not experience a relapse prior to discontinuation. Probability of participants who were relapse free at Year 3, estimated using the KM method, was reported.
Time Frame: Year 3
Population: FAS population included all randomized participants who had correct diagnosis of MS at entry.
Measure: Number (95% Confidence Interval); unit: probability of participants
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Alemtuzumab (Pooled)
Number analyzed (Participants) | 111 | 112 | 110 | 222
probability of participants | 0.50 [0.395 to 0.602] | 0.76 [0.667 to 0.832] | 0.84 [0.748 to 0.894] | 0.80 [0.737 to 0.847]
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Cox PH regression model with treatment group indicator, Baseline EDSS and country as covariates was used; Test type: Superiority or Other; p = 0.0001, Cox Proportional Hazards Regression; Treatment effect = 62.64
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Alemtuzumab 24 mg; Cox PH regression model with treatment group indicator, Baseline EDSS and country as covariates was used; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazards Regression; Treatment effect = 76.71
Statistical Analysis 3: Comparison: Interferon Beta-1a vs Alemtuzumab (Pooled); Cox PH regression model with treatment group indicator, Baseline EDSS and country as covariates was used; Test type: Superiority or Other; p < 0.0001, Cox Proportional Hazards Regression; Treatment effect = 70.13

4. Secondary Outcome: Percent Change From Baseline in T1 Cerebral Volume at Year 3
Description: Magnetic resonance imaging (MRI) T1 was used to determine rate of cerebral atrophy (decrease in cerebral/brain volume). Partial brain volumes were measured using the technique of Losseff et al. (1996). Percent change in cerebral volume at Year 3 was calculated from MRI-T1-weighted scans as: 100*([brain volume at Year 3] minus [brain volume at Baseline]) divided by [brain volume at Baseline]).
Time Frame: Baseline, Year 3
Population: Analysis population included participants in the FAS population (randomized with a correct diagnosis of MS) who had an evaluable scan for MRI-T1 brain volume at Baseline and Year 3.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Alemtuzumab (Pooled)
Number analyzed (Participants) | 67 | 83 | 90 | 173
percent change | -1.9 (4.48) | -0.8 (3.66) | -0.4 (4.27) | -0.6 (3.99)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Ranked analysis of covariance (ANCOVA) model using Baseline MRI-T1 brain volume, EDSS group, country, and treatment as covariates was used; Test type: Superiority or Other; p = 0.0885, ANCOVA
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Alemtuzumab 24 mg; Ranked ANCOVA model using Baseline MRI-T1 brain volume, EDSS group, country, and treatment as covariates was used; Test type: Superiority or Other; p = 0.0195, ANCOVA
Statistical Analysis 3: Comparison: Interferon Beta-1a vs Alemtuzumab (Pooled); Ranked ANCOVA model using Baseline MRI-T1 brain volume, EDSS group, country, and treatment as covariates was used; Test type: Superiority or Other; p = 0.0215, ANCOVA

5. Secondary Outcome: Percent Change From Baseline in MRI T2 Lesion Volume at Year 3
Description: Percent change in lesion volume at Year 3 was calculated from MRI-T2-weighted scans as: 100*([lesion volume at Year 3] minus [lesion volume at Baseline]) divided by [lesion volume at Baseline]).
Time Frame: Baseline, Year 3
Population: Analysis population included participants in the FAS population (randomized with a correct diagnosis of MS) who had an evaluable scan for MRI-T2 lesion volume at Baseline and Year 3.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Alemtuzumab (Pooled)
Number analyzed (Participants) | 66 | 81 | 88 | 169
percent change | 23.4 (134.3) | -11.4 (38.8) | -8.9 (41.1) | -10.1 (39.9)
Statistical Analysis 1: Comparison: Interferon Beta-1a vs Alemtuzumab 12 mg; Ranked ANCOVA model using Baseline MRI-T2 lesion volume, EDSS group, country, and treatment as covariates was used; Test type: Superiority or Other; p = 0.3077, ANCOVA
Statistical Analysis 2: Comparison: Interferon Beta-1a vs Alemtuzumab 24 mg; Ranked ANCOVA model using Baseline MRI-T2 lesion volume, EDSS group, country, and treatment as covariates was used; Test type: Superiority or Other; p = 0.3632, ANCOVA
Statistical Analysis 3: Comparison: Interferon Beta-1a vs Alemtuzumab (Pooled); Ranked ANCOVA model using Baseline MRI-T2 lesion volume, EDSS group, country, and treatment as covariates was used; Test type: Superiority or Other; p = 0.2758, ANCOVA

ADVERSE EVENTS:
Time Frame: First dose of study drug up to last follow-up (80.6 months)
Description: If a participant experienced both a serious and a non-serious event with the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables. The analysis was performed on the safety population, defined as all participants who received any amount of study drug.
Arm/Group | Interferon Beta-1a | Alemtuzumab 12 mg | Alemtuzumab 24 mg | Alemtuzumab (Pooled)
Serious Adverse Events (participants affected / at risk) | 29/107 | 30/108 | 33/108 | 63/216
Other Adverse Events (participants affected / at risk) | 106/107 | 108/108 | 108/108 | 216/216
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=107) | Alemtuzumab 12 mg (N=108) | Alemtuzumab 24 mg (N=108) | Alemtuzumab (Pooled) (N=216)
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 0 | 1
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 0 | 2 | 2
Thyroiditis subacute (Endocrine disorders) | 0 | 0 | 1 | 1
Cataract (Eye disorders) | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Exophthalmos (Eye disorders) | 0 | 1 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 1
Visual acuity reduced (Eye disorders) | 0 | 1 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Salivary gland calculus (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 1
Death (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Catheter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis of male external genital organ (Infections and infestations) | 0 | 0 | 1 | 1
Cervicitis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 2
Herpes ophthalmic (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis listeria (Infections and infestations) | 0 | 0 | 1 | 1
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Varicella (Infections and infestations) | 0 | 1 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic lung injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Ataxia (Nervous system disorders) | 2 | 0 | 1 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 2 | 2
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebellar ataxia (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1 | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 1 | 1
Multiple sclerosis relapse (Nervous system disorders) | 14 | 5 | 9 | 14
Myelitis (Nervous system disorders) | 0 | 1 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1 | 1
Paresis (Nervous system disorders) | 0 | 1 | 0 | 1
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0 | 0
Sensory loss (Nervous system disorders) | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 1 | 2
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 2 | 2
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 1
Goodpasture's syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 2 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Ectropion of cervix (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Interferon Beta-1a (N=107) | Alemtuzumab 12 mg (N=108) | Alemtuzumab 24 mg (N=108) | Alemtuzumab (Pooled) (N=216)
Neutropenia (Blood and lymphatic system disorders) | 1 | 6 | 4 | 10
Palpitations (Cardiac disorders) | 3 | 6 | 8 | 14
Tachycardia (Cardiac disorders) | 6 | 13 | 13 | 26
Vertigo (Ear and labyrinth disorders) | 10 | 12 | 11 | 23
Basedow's disease (Endocrine disorders) | 1 | 12 | 6 | 18
Hyperthyroidism (Endocrine disorders) | 1 | 11 | 13 | 24
Hypothyroidism (Endocrine disorders) | 1 | 11 | 11 | 22
Diplopia (Eye disorders) | 7 | 3 | 6 | 9
Vision blurred (Eye disorders) | 4 | 9 | 16 | 25
Visual acuity reduced (Eye disorders) | 6 | 4 | 2 | 6
Abdominal pain (Gastrointestinal disorders) | 7 | 6 | 5 | 11
Abdominal pain upper (Gastrointestinal disorders) | 6 | 2 | 4 | 6
Constipation (Gastrointestinal disorders) | 9 | 9 | 6 | 15
Diarrhoea (Gastrointestinal disorders) | 7 | 17 | 17 | 34
Dyspepsia (Gastrointestinal disorders) | 9 | 16 | 13 | 29
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 6 | 7 | 13
Nausea (Gastrointestinal disorders) | 17 | 32 | 45 | 77
Stomatitis (Gastrointestinal disorders) | 1 | 2 | 9 | 11
Toothache (Gastrointestinal disorders) | 1 | 1 | 6 | 7
Vomiting (Gastrointestinal disorders) | 9 | 18 | 19 | 37
Asthenia (General disorders) | 5 | 18 | 12 | 30
Chest discomfort (General disorders) | 3 | 12 | 18 | 30
Chills (General disorders) | 8 | 19 | 21 | 40
Fatigue (General disorders) | 31 | 47 | 44 | 91
Gait disturbance (General disorders) | 13 | 6 | 5 | 11
Hyperthermia (General disorders) | 1 | 7 | 5 | 12
Influenza like illness (General disorders) | 32 | 21 | 15 | 36
Injection site erythema (General disorders) | 35 | 1 | 0 | 1
Injection site pain (General disorders) | 18 | 3 | 0 | 3
Injection site reaction (General disorders) | 12 | 1 | 0 | 1
Oedema peripheral (General disorders) | 4 | 6 | 3 | 9
Pain (General disorders) | 6 | 13 | 14 | 27
Pyrexia (General disorders) | 11 | 47 | 47 | 94
Bronchitis (Infections and infestations) | 3 | 11 | 14 | 25
Herpes zoster (Infections and infestations) | 1 | 4 | 8 | 12
Influenza (Infections and infestations) | 4 | 10 | 3 | 13
Nasopharyngitis (Infections and infestations) | 14 | 17 | 26 | 43
Oral herpes (Infections and infestations) | 1 | 7 | 8 | 15
Pharyngitis (Infections and infestations) | 4 | 3 | 9 | 12
Rhinitis (Infections and infestations) | 3 | 9 | 9 | 18
Sinusitis (Infections and infestations) | 9 | 13 | 18 | 31
Upper respiratory tract infection (Infections and infestations) | 10 | 21 | 28 | 49
Urinary tract infection (Infections and infestations) | 11 | 11 | 17 | 28
Viral infection (Infections and infestations) | 6 | 4 | 2 | 6
Contusion (Injury, poisoning and procedural complications) | 3 | 6 | 15 | 21
Alanine aminotransferase increased (Investigations) | 9 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 6 | 7
Weight decreased (Investigations) | 2 | 7 | 9 | 16
Weight increased (Investigations) | 7 | 9 | 11 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 21 | 11 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 17 | 27 | 44
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 | 19 | 20 | 39
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 7 | 2 | 9
Muscular weakness (Musculoskeletal and connective tissue disorders) | 30 | 17 | 20 | 37
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9 | 10 | 5 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 11 | 12 | 23
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 7 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 25 | 32 | 57
Ataxia (Nervous system disorders) | 13 | 5 | 3 | 8
Balance disorder (Nervous system disorders) | 5 | 7 | 5 | 12
Burning sensation (Nervous system disorders) | 5 | 2 | 8 | 10
Coordination abnormal (Nervous system disorders) | 6 | 6 | 4 | 10
Dizziness (Nervous system disorders) | 11 | 13 | 29 | 42
Dysgeusia (Nervous system disorders) | 22 | 18 | 19 | 37
Headache (Nervous system disorders) | 26 | 72 | 85 | 157
Hypoaesthesia (Nervous system disorders) | 24 | 29 | 26 | 55
Migraine (Nervous system disorders) | 4 | 9 | 6 | 15
Multiple sclerosis (Nervous system disorders) | 5 | 8 | 6 | 14
Multiple sclerosis relapse (Nervous system disorders) | 40 | 27 | 21 | 48
Muscle spasticity (Nervous system disorders) | 8 | 4 | 0 | 4
Paraesthesia (Nervous system disorders) | 18 | 36 | 22 | 58
Sensory disturbance (Nervous system disorders) | 8 | 7 | 7 | 14
Tremor (Nervous system disorders) | 5 | 7 | 6 | 13
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 9 | 11 | 6 | 17
Anxiety (Psychiatric disorders) | 10 | 12 | 20 | 32
Depression (Psychiatric disorders) | 20 | 19 | 18 | 37
Insomnia (Psychiatric disorders) | 17 | 36 | 29 | 65
Micturition urgency (Renal and urinary disorders) | 6 | 1 | 6 | 7
Pollakiuria (Renal and urinary disorders) | 6 | 4 | 6 | 10
Urinary incontinence (Renal and urinary disorders) | 6 | 6 | 3 | 9
Urinary retention (Renal and urinary disorders) | 6 | 0 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 12 | 12 | 24
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 17 | 18 | 35
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 7 | 6 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 16 | 14 | 30
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 6 | 7 | 13
Erythema (Skin and subcutaneous tissue disorders) | 5 | 10 | 8 | 18
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 2 | 6 | 5 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 36 | 28 | 64
Rash (Skin and subcutaneous tissue disorders) | 8 | 78 | 82 | 160
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 13 | 7 | 20
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 6 | 4 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 3 | 31 | 38 | 69
Flushing (Vascular disorders) | 6 | 12 | 8 | 20
Hypertension (Vascular disorders) | 8 | 6 | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after sponsor publishes or 18 months after study completion. PI gives sponsor a draft 60 days before publication. Sponsor can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.